CLINICAL TRIAL: NCT05960396
Title: Exploring the Mechanism of Dietary Pattern Improving MAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230683
Record Dates: First submitted 2023-07-06; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: NAFLD; Diet Habit
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balanced diet (Experimental): Carbohydrates 50% -65%, fats 20% -30%, and proteins 10% -15%.
  Interventions: Behavioral: Diet intervention
- Low-carbohydrate diet (Experimental): Carbohydrates 20% -40%, fats 30% -45%, and proteins 30% -40%.
  Interventions: Behavioral: Diet intervention

INTERVENTIONS:
Behavioral: Diet intervention — investigators use different diet intervention to observe the changes of biochemical indicators, body composition, Gut microbiota, metabonomics, etc. for patients with MAFLD during different periods

SUMMARY:
investigators plan to observe the changes of biochemical indicators, body composition, gut microbiota, metabolomics in patients at different periods through balanced diet and Low-carbohydrate diet, so as to determine the beneficial "intestinal functional group" of MAFLD, and provide basis for the selection of the best time for probiotics and fecal bacteria transplantation.By comparing the response of the main outcome indicators to the two dietary structures, personalized nutritional intervention measures can be achieved.

DETAILED DESCRIPTION:
1. Balanced diet group: carbohydrates 50% -65%, fats 20% -30%, and proteins 10% -15%, among which proteins mainly come from beans, soy products, nuts, milk, poultry meat, aquatic products, and animal meat (lean); Lipids mainly come from Unsaturated fat acids, reducing the intake of Saturated fat acids; Carbohydrates mainly come from staple foods, with a combination of coarse and fine staple foods；
2. Low-carbohydrate diet intervention : carbohydrate 20% -40%, fat 30% -45%, protein 30% -40%. The protein mainly comes from beans, soy products, nuts, milk, meat, etc; Lipids mainly come from Unsaturated fat acids, reducing the intake of Saturated fat acids; Carbohydrates mainly come from low GI foods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old, Han nationality, residing in China ；

  * MRI-PDFF ≥ 5% or /and control attenuation index (CAP value) ≥ 244db /m and Alanine transaminase or /and cereal grass Transaminase are within 3 times of the upper limit of normal value;

    * At least one metabolic disease exists: BMI ≥ 24kg/m2; According to widely recognized international standards, it is diagnosed as type 2 diabetes [diabetes symptoms+plasma glucose level at any time ≥ 200mg /dl (11.1mmol /L) or fasting plasma glucose ≥ 126mg /dl (7.0mmol /L) or in Oral Glucose Tolerance Test test, blood glucose at 2 hours after meal ≥ 200mg /dl (11.1mmol /L)]; There are at least two risk factors for metabolic abnormalities: a Waist circumference: male ≥ 90cm, female ≥ 80cm; B Blood pressure ≥ 130/85mmHg or receiving specific drug treatment; C Plasma triglycerides ≥ 150mg/dl (≥ 1.70mmol/L) or receiving specific drug treatment; D Plasma High-density lipoprotein cholesterol: male<40mg /dl (<1.0mmol /L) and female<50mg /dl (<1.3mmol /L) or receive specific drug treatment; E Pre diabetes [i.e. Glucose test#Fasting blood sugar level is 100~125mg /dl (5.6~6.9 mmol /L), or blood glucose level 2 hours after meal is 140~199mg /dl (7.8~11.0 mmol /L) or Glycated hemoglobin is 5.7%~6.4% (39~47 mmol /L)]; F steady-state model evaluation - insulin resistance index ≥ 2.5; The plasma level of hypersensitive C-reactive protein is ≥ 2mg/L.

      * Willing to accept evaluation and sign informed consent

Exclusion Criteria:

* Fatty liver patients undergoing medication treatment;

  * Those who have received weight loss treatment such as medication, surgery, or meal replacement within the past 3 months;

    * Those who currently or in the past 3 weeks have taken antibiotics, probiotics, prebiotics or other microbiota related supplements;

      * Receive Corticosteroid or Thyroid hormones treatment; ⑤ Having clinically diagnosed viral hepatitis, autoimmune liver disease, cirrhosis and other liver diseases

        * Secondary obesity caused by endocrine, genetic, metabolic and Central nervous system disease; ⑦ Patients with abnormal liver function (Alanine transaminase or /and glutamic oxalic Transaminase exceed the upper limit of normal value by 3 times); Patients with renal dysfunction (serum creatinine exceeding the upper limit of normal values); Suffering from diseases such as kidney disease that require protein intake control;

          * Diseases affecting food digestion and absorption (such as chronic diarrhea, constipation, severe gastrointestinal inflammation, active gastrointestinal ulcer, postoperative gastrointestinal tract resection, Cholecystitis /cholecystectomy, etc.); ⑨ Suffering from cardio cerebral Vascular disease, grade 3 hypertension, chronic hepatitis, malignant tumor, anemia, mental disease, memory impairment, epilepsy and other diseases ⑩ having major diseases or having recently undergone Major trauma /surgery, etc

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
changes of liver fat content before and after interventions | 0month and 12month
  Measurement of liver fat content was undertaken at baseline and at the end of the study by using proton magnetic resonance spectroscopy (MRS)

CONTACTS AND LOCATIONS:
Overall Officials: the second affiliated hospital of zhejiang university, Principal Investigator — Zhejiang University

IPD SHARING:
Plan to Share IPD: No